CLINICAL TRIAL: NCT00583635
Title: Minimizing Early Pregnancy Oxidative Stress to Maximize Healthy Pregnancy Outcome: Reducing Preeclampsia and Reproductive Loss With Antioxidant-Rich Tablet Supplementation Initiated in the First Trimester
Brief Title: Early Pregnancy Antioxidant Supplementation in the Prevention of Preeclampsia
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, James Martin, Professor, University of Mississippi Medical Center
Other Study IDs: IRB File # 2003-0119
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Preeclampsia; Pregnancy Loss
Keywords: Preeclampsia; Prevention; Food Supplement
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood to be analyzed for various markers, then discarded, none to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Low Risk Pregnancy, Placebo
- 2: Low Risk Pregnancy, Active Food Supplement
- 3: High Risk Pregnancy, Placebo
- 4: High Risk Pregnancy, Active Food Supplement

SUMMARY:
Use of Juice Plus+ food supplements, when initiated in the first trimester and used continuously thereafter, will result in a lower incidence of preeclampsia and pregnancy complications. This is a prospective randomized and blinded placebo controlled study sponsored by NSA, LLC of Memphis, TN.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Patients seen in first trimester with low or high risk pregnancy

Exclusion Criteria:

* Pregnant patients first seen after the first trimester
* Unlikely to continue care in our system
* Unwilling to comply with rigor of taking food supplements throughout gestation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients cared for in the University of Mississippi Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2004-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Development of preeclampsia during pregnancy | Preeclampsia at any time during gestation

SECONDARY OUTCOMES:
The observed incidence of preterm labor, premature rupture of membranes, perinatal loss | First, second and third trimester

CONTACTS AND LOCATIONS:
Overall Officials: James N Martin, Jr., MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States